CLINICAL TRIAL: NCT01997944
Title: Phase Ib Study of Recombinant Human Serum Albumin/Interferon alpha2a Fusion Protein in Chronic Hepatitis B Patients
Brief Title: Recombinant Human Serum Albumin/Interferon alpha2a Fusion Protein Phase Ib Study in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Bio-Fortune Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 921302
Record Dates: First submitted 2013-11-21; First posted 2013-11-28 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Serum Albumin, Human; Interferon alpha-2; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Serum Albumin/interferon alpha2a (Experimental): Human Serum Albumin/interferon alpha2a 600,750 or 900 mcg multiple dose S.C.
  Interventions: Biological: Human Serum ALbumin/interferon alpha2a
- Pegasys (Active Comparator): Peginteferon 180 mcg multiple dose S.C.
  Interventions: Biological: Pegasys

INTERVENTIONS:
Biological: Human Serum ALbumin/interferon alpha2a — 600,750 or 900 mcg dosing every 2 weeks
  Arms: Human Serum Albumin/interferon alpha2a
Biological: Pegasys — 180 mcg dosing every week
  Arms: Pegasys

SUMMARY:
This is an open label study that will be conducted at a single site in China to evaluate the safety,tolerability and PK/PD profile of multiple dose of recombinant human serum albumin/interferon alpha2a fusion protein in chronic hepatitis B patients.The total duration of study participation is up to 22 weeks for each subject,including 4 weeks screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years
* Chronic HBV infection (serum HBsAg detectable for > 6 months)
* Serum HBeAg positive with HBV DNA >10^6copies/mL (or >20,000 IU/mL),orSerum HBeAg negative with HBV DNA >10^5copies/mL (or >2,000 IU/mL)
* Serum ALT must be > 2 x ULN but below 10 x ULN

Exclusion Criteria:

* Steroid treatment or immunosuppression 3 months prior to entry.
* Interferon therapy or nucleotides analogues therapy in 6 months prior to entry.
* Active lung disease or history of interstitial lung disease.
* Hb< LLN or, and ANC < 750/mm3 or , and platelet count < 75,000 mm3 ,or WBC<3000/mm3 .
* Significant chronic medical conditions other than chronic hepatitis B which in the opinion of the investigator preclude enrollment into the study.
* Evidence of hepatic decompensation (i.e., Child-Pugh score of B or C).
* Seropositive for HIV, HCV, or HDV (Hepatitis Delta virus).
* History of thyroid disease or current treatment for thyroid disease.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 18 weeks

SECONDARY OUTCOMES:
Decrease of HBV DNA | 18 weeks
AUCss | 18 weeks
Css_av | 18 weeks
Css_min | 18 weeks
Css-max | 18 weeks
T1/2 | 18 weeks
Tmax | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, MD, Principal Investigator — Jilin University First Affiliated Hospital
Locations (1):
- Jilin University First Affiliated Hospital, Changchun, Jilin, China